CLINICAL TRIAL: NCT02496390
Title: Transplantation of Microbes of Fecal Origin for Prevention and Treatment of Metabolic Syndrome and Non Alcoholic Fatty Liver Disease
Brief Title: Transplantation of Microbes for Treatment of Metabolic Syndrome & NAFLD
Acronym: FMT
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IDFMT - 001
Record Dates: First submitted 2015-07-07; First posted 2015-07-14 (Estimated); Last update posted 2018-12-11 (Actual); Status verified 2018-12

CONDITIONS: Diabetes Mellitus; Non-alcoholic Fatty Liver Disease
Keywords: Fecal Microbial Transplantation; Gut microbiome; Metabolic disorders; Obesity
MeSH Terms: conditions — Diabetes Mellitus; Non-alcoholic Fatty Liver Disease; Metabolic Diseases; Obesity

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Autologous (Placebo Comparator): Patients will be randomized to receive a fecal transplant using their own microbes/Feces (autologous - 9 patients).
  Dosage - approx 100ml fecal sample, one time, procedure duration ~1hr
  Interventions: Biological: Autologous
- Allogenic (Active Comparator): Patients will be randomized to receive a fecal transplant of feces/microbiome from the healthy donor (allogeneic - 12 patients).
  Dosage - approx 100ml fecal sample, one time, procedure duration ~1hr
  Interventions: Biological: Allogeneic

INTERVENTIONS:
Biological: Autologous — Patients will have their normal microbiome reduced using an oral preparation (pico-salax) as used for routine colonic preparation for colonoscopy. • Administration of the FMT will be via a nasoduodenal tube inserted at the time of gastroscopy. Dosage - approx 100ml previously frozen fecal sample obtained from the patient prior to colonic preparation.
  Other Names: Autologous fecal infusions
  Arms: Autologous
Biological: Allogeneic — Patients will have their normal microbiome reduced using an oral preparation (pico-salax) as used for routine colonic preparation for colonoscopy. • Administration of the FMT will be via a nasoduodenal tube inserted at the time of gastroscopy. Dosage - approx 100ml previously frozen fecal sample obtained from a lean donor prior to colonic preparation.
  Other Names: Fecal Microbial Transplantation
  Arms: Allogenic

SUMMARY:
Non-alcoholic fatty liver disease (NAFLD) occurs when excess fat is deposited in the liver. Almost all patients also have obesity and insulin resistance (the inability of the body to effectively use insulin). Obesity and NAFLD are intricately intertwined and are increasing in incidence. While weight loss is the most effective therapy for NAFLD, the investigators' efforts are failing and in the next generation it will become the most common cause of liver failure in Canada. Recently, researchers have focused on the potential use of altering the composition of bacteria in the gut (microbiome) to alter absorption of energy from food, deposition of fat and resistance to insulin. This study will determine if transplantation of bacteria from the stool of a healthy volunteer into an individual with metabolic syndrome and NAFLD (i.e. fecal microbiota transplant/FMT) can alter insulin resistance and reduce the amount of fat deposited in the liver. FMT is being studied to treat several clinical conditions and is now standard of care for the treatment of refractory Clostridium difficile infection. Investigators are proposing a randomized controlled pilot study of FMT in 21 patients to determine the feasibility and to inform us of changes needed for a larger study.

DETAILED DESCRIPTION:
Obesity and obesity-related disorders such as metabolic syndrome, Type 2 Diabetes (DM2), and NAFLD are of increasing concern worldwide. Metabolic syndrome refers to the clustering of 3 out of 5 parameters - abdominal obesity, elevated blood pressure, elevated fasting glucose, elevated triglyceride level, and low high-density lipoprotein cholesterol (HDL-C) level. The prevalence of metabolic syndrome is approximately 20-25% in North America. Those with metabolic syndrome are at increased risk for DM2 and cardiovascular disease.

Metabolic syndrome, DM2 and NAFLD are all marked by insulin resistance and are intricately linked with obesity. NAFLD is currently the most common liver disease in developed countries such as Canada. About 10-20% of patients with NAFLD progress to non-alcoholic steatohepatitis (NASH) which is characterized by inflammation and fat deposition. Unfortunately, NASH is a major cause of cirrhosis in North America.

Gut Microbiota, Obesity, DM2, and NAFLD Very strong support for the hypothesis of the gut microbiome inducing insulin resistance was found in a recent randomized control trial which showed that fecal transplantation from lean healthy donors into human patients with metabolic syndrome resulted in improved insulin sensitivity. This improvement correlated to an increase in the prevalence of butyrate-producing bacteria. Since butyrate helps prevent programmed cell death in the mucosal cells of the colon, preserving the integrity of the intestinal mucosa may prevent migration of endotoxin from the gut to the liver and induction of insulin resistance. Larger metagenome wide association studies of the fecal microbiome confirmed this finding that butyrate-producing bacteria including Clostridiales spp,C. rectales, Faecalibacterium prausnitzii, Roseburia intestinalis and R.inulinvorans appear to be less prevalent in DM2 than in healthy controls.

Differences in the microbiome between obese patients and those with DM2 versus those with a normal body mass index have been reported in many publications. There is evidence that the altered flora can increase the efficiency of release of calories from food. In a study of obese human twins, the decrease in Bacteroidetes proportion with increase in Firmicutes proportion correlated with the enrichment of microbial genes encoding key enzymes involved in carbohydrate metabolism, potentially leading to increased digestion of food and supply of energy in the form of short chain fatty acids (SCFA) to the host. Transfer of the gut microbiota from obese mice or from obese humans into germ-free mice reproduced the obese phenotype. Differences in microbiota composition have even been documented between children with obesity and those children who are lean, suggesting that microbiota changes may occur early in life. Decrease in the ratio of the number of firmicutes/bacteroidetes were associated with weight loss in humans. Other human gut organisms such as Akkermansia muciniphilia and Enterobacter cloacae B29 have been implicated with obesity and DM2. A high concentration of gut Beta proteobacteria was associated with the development of diabetes possibly via an inflammatory response incited by the endotoxin within these Gram negative rods. In fact antibiotic administration in some animal models has led to reduced numbers of both aerobic and anaerobic bacteria which increases insulin sensitivity as well as in plasma adiponectin levels, which correlate with insulin sensitivity. Changes in the gut microbiota associated with obesity have been found to activate Toll like receptors and thus GI inflammation with resulting insulin resistance. Very recently it was found that artificial sweeteners despite being "no-calorie" can exacerbate glucose intolerance, the effect mediated via a change in the microbiome.

Compared to both healthy controls and simple steatosis patients, patients with NASH have a lower percentage of the phylum Bacteroidetes, a finding similar to that of the gut microbial flora in obese human subjects. Microbial fermentation products like ethanol in the gut are key factors to induce obesity in mice and may be related to the pathogenesis of fatty liver disease. Elevated systemic ethanol levels even in the absence of any ethanol ingestion have been noted in patients with NASH compared to controls, suggesting that ethanol-producing microbes might be related to the pathogenesis of NASH in humans.Certain microbiomes can also lead to higher monosaccharide absorption from the gut lumen, which can promote de novo fatty acid and triglyceride production in the liver. It has been found that the hepatic kupffer cell activation in mice seems to contribute to the pathogenesis of NAFLD and that this can be induced by microbial endotoxin-related chronic inflammation. Chronic endotoxemia is associated with the severity of NAFLD. Increased intestinal permeability has similarly been documented in DM2 and metabolic syndrome and likely plays a key role in the pathophysiology of these disorders. Overall these findings suggest that preventive or therapeutic interventions such as fecal transplantation may lead to improvement in the status of obesity, metabolic syndromes, and NASH or NAFLD,and possibly even atherosclerosis.

Fecal Microbial Transplantation has been used extensively in humans with recurrent C.difficile infection and has been found to be safe, effective and well tolerated. Frozen stool has been found to be equally safe and effective to fresh stool for transplant. This procedure has become well accepted and is now considered the standard of practice for patients with recurrent C.difficile, and is included in newer practice guidelines. Its use in metabolic syndromes is new, but the safety data from the much larger experience in patients with C.difficile is very reassuring.

Goal:

• To determine the impact of alterations of the gut microbiome on parameters of insulin resistance and on liver fat content.

Rationale:

As mentioned in the background review there is extensive animal and also moderately extensive human studies demonstrating that alteration in the microbiome is associated with metabolic syndrome and NAFLD. There is also extensive biochemical rationale for why microbiome changes could lead to the changes in the metabolic outcomes in humans.

Justification of Innovation:

The inability of existing therapies to control weight gain, obesity and associated liver diseases in individuals with metabolic disorders is a major public health concern. The potential of gut microbial alteration to prevent and control metabolic disorders (duplicating the success of FMT for Clostridium difficile infection) would be an important advance. This will be a proof of concept study which will enable further more targeted innovations of the gut microbiome to control the metabolic syndrome and NAFLD.

ELIGIBILITY:
* Gender: Male: only male participants are being studied
* Age limits: Minimum - 18yrs and above and Maximum-NA
* Eligibility Criteria: Participants who meet the criteria's mentioned below will only be selected for the study
* Inclusion Criteria:
* Attendance at the gastroenterology/hepatology clinic with a diagnosis of NAFLD as well as metabolic syndrome.
* Ability to provide informed Consent.
* Exclusion Criteria:
* Type 1 or 2 Diabetes requiring ongoing hypoglycemic medications.
* Inability to attend follow-up visits.
* Inability to provide informed written consent.
* Ongoing use of antibiotics or probiotics.
* Previous or planned bariatric surgery.
* Presence of a chronic intestinal disease e.g. Celiac, malabsorption, Colonic tumor.
* Immunosuppression from transplantation, HIV, Cancer chemotherapy or ongoing use of any immunosupressive agents.
* Pregnant women
* Any contra-indications for MRI as listed below: a. Previous brain surgery (using the language outlined in the Health Sciences Research Ethics Board [HSREB] Guideline, section 2-G-004) Pacemaker, Cerebral aneurism clips, neurostimulator, Metallic heart valves, Intra Uterine Devices [IUD], Joint replacement, Metal plates Bone or joint pins, Venacava filters, Embolization coils, Cochlear implants, Greenfield Filter, Seizures, Claustrophobia, Bullet/gunshot wound, Non-removable prosthesis, Non-removable artificial limbs, Surgical clips, Metal screws or pins, Shrapnel/metallic fragments, Harrington rod, Insulin pump, Ever had metal removed from in or around the eye, Ever been a metal worker (i.e. welder, machinist), Non-removable hearing aids, Bird nest or Gianturco filter, Metal braces, Severe heart disease (including susceptibility to arrhythmias), Weight or body habitus that will prevent a successful MRI study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2018-04 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Improvement in Homeostasis model assessment [HOMA] score. | 6 weeks

SECONDARY OUTCOMES:
Fat reduction | 6 months
  Percentage of fat in liver Magnetic Resonance Imaging [MRI]
Reducing body fat | 6 months
  Change in waist circumference and weight
Gut permeability | 6 months
  Change in percentage lactulose absorption
Microbiome modulation | 6 months
  Change in microbiome of stool and duration of change before reverting to baseline
Modulation of lipid and hormone metabolism | 6 months
  Change in markers of lipid metabolism and hormones associated with adiposity

CONTACTS AND LOCATIONS:
Overall Officials: Michael Silverman, MD, Principal Investigator — London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Locations (1):
- Michael Silverman, London, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vrieze A, Van Nood E, Holleman F, Salojarvi J, Kootte RS, Bartelsman JF, Dallinga-Thie GM, Ackermans MT, Serlie MJ, Oozeer R, Derrien M, Druesne A, Van Hylckama Vlieg JE, Bloks VW, Groen AK, Heilig HG, Zoetendal EG, Stroes ES, de Vos WM, Hoekstra JB, Nieuwdorp M. Transfer of intestinal microbiota from lean donors increases insulin sensitivity in individuals with metabolic syndrome. Gastroenterology. 2012 Oct;143(4):913-6.e7. doi: 10.1053/j.gastro.2012.06.031. Epub 2012 Jun 20. PMID 22728514
- [Background] van Nood E, Vrieze A, Nieuwdorp M, Fuentes S, Zoetendal EG, de Vos WM, Visser CE, Kuijper EJ, Bartelsman JF, Tijssen JG, Speelman P, Dijkgraaf MG, Keller JJ. Duodenal infusion of donor feces for recurrent Clostridium difficile. N Engl J Med. 2013 Jan 31;368(5):407-15. doi: 10.1056/NEJMoa1205037. Epub 2013 Jan 16. PMID 23323867
- [Background] Hamilton MJ, Weingarden AR, Sadowsky MJ, Khoruts A. Standardized frozen preparation for transplantation of fecal microbiota for recurrent Clostridium difficile infection. Am J Gastroenterol. 2012 May;107(5):761-7. doi: 10.1038/ajg.2011.482. Epub 2012 Jan 31. PMID 22290405
- [Background] Kunde S, Pham A, Bonczyk S, Crumb T, Duba M, Conrad H Jr, Cloney D, Kugathasan S. Safety, tolerability, and clinical response after fecal transplantation in children and young adults with ulcerative colitis. J Pediatr Gastroenterol Nutr. 2013 Jun;56(6):597-601. doi: 10.1097/MPG.0b013e318292fa0d. PMID 23542823
- [Background] Bailey LC, Forrest CB, Zhang P, Richards TM, Livshits A, DeRusso PA. Association of antibiotics in infancy with early childhood obesity. JAMA Pediatr. 2014 Nov;168(11):1063-9. doi: 10.1001/jamapediatrics.2014.1539. PMID 25265089
- [Derived] Aghara H, Patel M, Chadha P, Parwani K, Chaturvedi R, Mandal P. Unraveling the Gut-Liver-Brain Axis: Microbiome, Inflammation, and Emerging Therapeutic Approaches. Mediators Inflamm. 2025 Jun 18;2025:6733477. doi: 10.1155/mi/6733477. eCollection 2025. PMID 40568349
- [Derived] Craven L, Rahman A, Nair Parvathy S, Beaton M, Silverman J, Qumosani K, Hramiak I, Hegele R, Joy T, Meddings J, Urquhart B, Harvie R, McKenzie C, Summers K, Reid G, Burton JP, Silverman M. Allogenic Fecal Microbiota Transplantation in Patients With Nonalcoholic Fatty Liver Disease Improves Abnormal Small Intestinal Permeability: A Randomized Control Trial. Am J Gastroenterol. 2020 Jul;115(7):1055-1065. doi: 10.14309/ajg.0000000000000661. PMID 32618656